CLINICAL TRIAL: NCT02360982
Title: Cukurova University Faculty of Medicine
Brief Title: The Comparison of Incidence and Risk Factors of Postoperative Delirium in Elderly Patients After Lower Extremity Surgery
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, specialist dr, Cukurova University
Other Study IDs: cukurova university
Record Dates: First submitted 2015-02-04; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Postoperative Delirium
Keywords: Delirium; regional anesthesia; general anesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Propofol; Bupivacaine; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- propofol and esmeron(rokuronyum): In group G, anesthesia was induced with iv propofol (2 mg.kg-1) and maintained with 2% sevoflurane in a mixture of 65 % nitrous oxide and 35 % oxygen with a total gas flow rate of 6 L min-1. Neuromuscular relaxation was induced with iv rocuronium (esmeron) (0.5 mg.kg-1). Intravenous infusion of 0.9% saline was administered at a volume of 5 mL/kg/h. Patients received morphine (0.1mg/kg) for postoperative analgesia 30 minutes before the end of the operation. Anesthesia was terminated and neuromuscular blockade was antagonized with neostigmine (0.05 mg.kg-1)and atropine sulphate (0.01 mg.kg-1).
  Interventions: Behavioral: propofol and esmeron(rokuronyum); Behavioral: marcaine and fentanyl
- marcaine and fentanyl: We inserted a 18-G Tuohy needle at the L3/L4 or L2/L3 intervertebral epidural space using an epidural loss of resistance technique and thus performed needle-through-needle technique for subarachnoid injection of 2 mL bupivacaine (marcaine)(0.5%) and fentanyl (25 mcg) by 27-G spinal needle. After subarachnoid injection, epidural catheter was advanced and fixed.
  At the end of the surgery 5 mL of bupivacaine 0.5% plus morphine (1 mg), adding to 4 mL saline was injected via epidural catheter for postoperative analgesia.Epidural catheter was removed at 24th hours
  Interventions: Behavioral: propofol and esmeron(rokuronyum); Behavioral: marcaine and fentanyl

INTERVENTIONS:
Behavioral: propofol and esmeron(rokuronyum) — All patients were evaluated at postoperative 24th and 72th hours with laboratory tests including hemoglobin, sodium, potassium, BUN, creatinine, total protein, albumin and glucose values in blood samples and delirium tests (CAM and DRS-R-98).
Behavioral: marcaine and fentanyl — All patients were evaluated at postoperative 24th and 72th hours with laboratory tests including hemoglobin, sodium, potassium, BUN, creatinine, total protein, albumin and glucose values in blood samples and delirium tests (CAM and DRS-R-98).

SUMMARY:
The aim of this study is to compare the risk factors and the incidence of delirium following orthopedic surgery under the general or regional anesthesia in elderly patients.

DETAILED DESCRIPTION:
One hundred twenty elderly patients aged ≥65 years scheduled for total hip or knee arthroplasty and femur fracture surgery were enrolled into the study. Patients were allocated into two groups to receive regional anesthesia (group R, n=50) or general anesthesia (group G, n=70). Hemodynamic and blood parameters, potential risk factors of delirium including age, sex, duration of surgery, the type of anesthesia, coexisting disease, smoking and amount of drug used delirium tests (CAM and DRS-R-98), hospital stay and costs were recorded for all patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-III,
* 120 patients aged ≥65 years scheduled for total hip or knee arthroplasty and femur fracture surgery

Exclusion Criteria:

* Exclusion criteria were patient refusal, abuse of alcohol and/or drugs
* Hypersensitivity to local anesthetics
* Vertebral abnormality
* Previous lumbar vertebra surgery
* Coagulation disorder
* Infection (systemic or local)
* Cerebrovascular disease
* Neurosurgery
* Vascular surgery
* Frequent use of analgesic drug
* ≥5 drugs per day and psychiatric medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: American Society of Anesthesiologists physical status I-III, 120 patients aged ≥65 years scheduled for total hip or knee arthroplasty and femur fracture surgery were enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
the presence of postoperative delirium as defined by CAM criteria. | one year

SECONDARY OUTCOMES:
severity of delirium rated with the DRS-R-9 | one year
length of hospital stay and costs. | one year

CONTACTS AND LOCATIONS:
Overall Officials: ILKE KUPELI, Principal Investigator — MENGUCEK GAZI TRAINING AND RESEARCH HOSPITAL DEPARTMENT OF ANESTHESIOLOGY AND INTENSIVE CARE; ERSEL GULEC, Study Chair — CUKUROVA UNIVERSITY DEPARTMENT OF ANESTHESIOLOGY AND INTENSIVE CARE; EBRU BIRICIK, Study Chair — CUKUROVA UNIVERSITY DEPARTMENT OF ANESTHESIOLOGY AND INTENSIVE CARE; AKIF MIRIOĞLU, Study Chair — CUKUROVA UNIVERSITY DEPARTMENT OF ORTHOPEDICS AND TRAUMATOLOGY; YASEMIN GUNES, Study Chair — CUKUROVA UNIVERSITY DEPARTMENT OF ANESTHESIOLOGY AND INTENSIVE CARE

REFERENCES:
- [Background] Litaker D, Locala J, Franco K, Bronson DL, Tannous Z. Preoperative risk factors for postoperative delirium. Gen Hosp Psychiatry. 2001 Mar-Apr;23(2):84-9. doi: 10.1016/s0163-8343(01)00117-7. PMID 11313076
- [Background] Schrader SL, Wellik KE, Demaerschalk BM, Caselli RJ, Woodruff BK, Wingerchuk DM. Adjunctive haloperidol prophylaxis reduces postoperative delirium severity and duration in at-risk elderly patients. Neurologist. 2008 Mar;14(2):134-7. doi: 10.1097/NRL.0b013e318166b88c. PMID 18332845
- [Background] Steiner LA. Postoperative delirium. Part 1: pathophysiology and risk factors. Eur J Anaesthesiol. 2011 Sep;28(9):628-36. doi: 10.1097/EJA.0b013e328349b7f5. PMID 21785356
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Bryson GL, Wyand A. Evidence-based clinical update: general anesthesia and the risk of delirium and postoperative cognitive dysfunction. Can J Anaesth. 2006 Jul;53(7):669-77. doi: 10.1007/BF03021625. PMID 16803914
- [Background] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- [Background] Papaioannou A, Fraidakis O, Michaloudis D, Balalis C, Askitopoulou H. The impact of the type of anaesthesia on cognitive status and delirium during the first postoperative days in elderly patients. Eur J Anaesthesiol. 2005 Jul;22(7):492-9. doi: 10.1017/s0265021505000840. PMID 16045136
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] Marcantonio E, Ta T, Duthie E, Resnick NM. Delirium severity and psychomotor types: their relationship with outcomes after hip fracture repair. J Am Geriatr Soc. 2002 May;50(5):850-7. doi: 10.1046/j.1532-5415.2002.50210.x. PMID 12028171
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695
- [Background] McAlpine JN, Hodgson EJ, Abramowitz S, Richman SM, Su Y, Kelly MG, Luther M, Baker L, Zelterman D, Rutherford TJ, Schwartz PE. The incidence and risk factors associated with postoperative delirium in geriatric patients undergoing surgery for suspected gynecologic malignancies. Gynecol Oncol. 2008 May;109(2):296-302. doi: 10.1016/j.ygyno.2008.02.016. Epub 2008 Mar 28. PMID 18374970
- [Background] Schuurmans MJ, Duursma SA, Shortridge-Baggett LM, Clevers GJ, Pel-Littel R. Elderly patients with a hip fracture: the risk for delirium. Appl Nurs Res. 2003 May;16(2):75-84. doi: 10.1016/s0897-1897(03)00012-0. PMID 12764718
- [Background] Martin NJ, Stones MJ, Young JE, Bedard M. Development of delirium: a prospective cohort study in a community hospital. Int Psychogeriatr. 2000 Mar;12(1):117-27. doi: 10.1017/s1041610200006244. PMID 10798458
- [Background] Radtke FM, Franck M, MacGuill M, Seeling M, Lutz A, Westhoff S, Neumann U, Wernecke KD, Spies CD. Duration of fluid fasting and choice of analgesic are modifiable factors for early postoperative delirium. Eur J Anaesthesiol. 2010 May;27(5):411-6. doi: 10.1097/EJA.0b013e3283335cee. PMID 19887950
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Rudolph JL, Jones RN, Levkoff SE, Rockett C, Inouye SK, Sellke FW, Khuri SF, Lipsitz LA, Ramlawi B, Levitsky S, Marcantonio ER. Derivation and validation of a preoperative prediction rule for delirium after cardiac surgery. Circulation. 2009 Jan 20;119(2):229-36. doi: 10.1161/CIRCULATIONAHA.108.795260. Epub 2008 Dec 31. PMID 19118253
- [Background] Elie M, Cole MG, Primeau FJ, Bellavance F. Delirium risk factors in elderly hospitalized patients. J Gen Intern Med. 1998 Mar;13(3):204-12. doi: 10.1046/j.1525-1497.1998.00047.x. PMID 9541379
- [Result] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989